CLINICAL TRIAL: NCT05323019
Title: A Randomized, Controlled, Single-Blind, Phase 2 Study in Treatment Resistant Major Depressive Disorder Patients Receiving Intranasal Esketamine (SpravatoTM) Over a 28-day Period Comparing Addition of Almond TherapyTM With Treatment-as-Usual
Brief Title: Repeated Intranasal Esketamine Plus Almond Therapy in Patients With Treatment Resistant Depression
Acronym: ZYL-730-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Zylorion Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA-CTC-22-0015
Record Dates: First submitted 2022-03-24; First posted 2022-04-12 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Treatment Resistant Major Depressive Disorder
MeSH Terms: interventions — Psychotherapy; Therapeutics; Esketamine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized by a pre-specified block design method after confirming eligibility.
Who Masked: Outcomes Assessor
Masking Description: The independent trained individual will not be aware of which treatment arm the participant has been randomized to. The MADRS assessor will have no other contact with the participants apart from remotely assessing the MADRS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal (esketamine) Ketamine with Addition of Almond therapy (Other): Intranasal (esketamine) Ketamine - Dose of 56mg for a maximum of 2 weeks, followed by 56 mg or 84mg twice a week for a total of 8 doses during the 28 day study.
  Interventions: Behavioral: Psychotherapy; Drug: Intranasal Ketamine (esketamine)
- Intranasal (esketamine) Ketamine with Treatment as Usual (Other): Intranasal (esketamine) Ketamine - Dose of 56 mg for a maximum of 2 weeks, followed by 56mg or 84mg twice a week for a total of 8 doses during the 28 day study.
  Interventions: Behavioral: Treatment as Usual; Drug: Intranasal Ketamine (esketamine)

INTERVENTIONS:
Behavioral: Psychotherapy — Participants will receive 8 remote therapy sessions conducted via phone or video, Therapy sessions consists of modules selected using a shared decision making process, tailored so that it is personally meaningful to each participant. Participants will also receive supportive text messages on selected days during the 28 day study.
  Arms: Intranasal (esketamine) Ketamine with Addition of Almond therapy
Behavioral: Treatment as Usual — Participants will continue to receive the therapy that their treating physician felt was appropriate at the time of enrolment in the study, These can include cognitive behavioural therapy, supportive psychotherapy or mindfulness, support groups, physical exercise or relaxation.
  Arms: Intranasal (esketamine) Ketamine with Treatment as Usual
Drug: Intranasal Ketamine (esketamine) — Intranasal Ketamine (esketamine) - participants will receive a dose of 56 mg for a maximum of 2 weeks, followed by 56 mg or 84 twice a week for a total of 8 doses during the 28 -day study
  Other Names: Spravato

SUMMARY:
To examine the efficacy of Almond Therapy compared to Treatment as Usual when used in addition to an approved version of intranasal esketamine.

DETAILED DESCRIPTION:
The duration of the study is 28 days.

Participants enrolled in the Almond Therapy arm will have up 10 in person clinic visits, including the screening visit, participants will receive esketamine on 8 of these visits. There are also 8 remote therapy sessions conducted via telephone or video, and participants will also receive supportive text messages. Participants will have 5 telephone calls from an independent assessor to ask questions about their mental health (MADRS).

Participants enrolled in the Treatment as usual will have 10 in-person clinic visits, including the Screening visit, participants will receive intranasal esketamine on 8 of these visits. Participants will continue to receive the therapy that their treating physician felt was appropriate at the time of enrolment in the study. In addition, participants will have 5 telephone calls from an independent assessor to ask questions on their mental health ( MADRS).

Participants will receive intranasal esketamine twice-weekly according to the Product Monograph. To ensure that both groups receive approximately equal amounts of esketamine, patients will receive 56mg initially for a maximum of 2 weeks followed by 56mg or 84mg. As per the Product Monograph these will be given for 4 weeks for a total of 8 doses during the 28-day study.

ELIGIBILITY:
Inclusion Criteria:

* Score on MADRS scale with a score of 18 or greater
* Meet criteria for Treatment-Resistant Major Depressive Disorder, defined as having not responded adequately to at least two separate courses of treatment with different antidepressant at an adequate dose and duration in the current moderate to severe depression episode, as determined by an appropriately trained psychiatrist.
* Women of child bearing potential must use a medically acceptable means of contraception for the duration of the study and for 6 weeks after the last dose of esktamine.
* Negative blood pregnancy test prior to baseline
* If currently receiving medication for depression, antidepressant dose must be stable for the previous 4 weeks prior to baseline.
* Stable dose of all other medication for at least 1 month prior to baseline
* Controlled hypertension and on a stable dose of antihypertension medications for at least 3 months prior to baseline visit

Exclusion Criteria:

* Women who plan to become pregnant, are pregnant or are breastfeeding
* Serious unstable medical illness as determined by the Investigator.
* Participants with uncontrolled hypothyroidism and hyperthyroidism
* Hormonal treatment (e.g., Estrogen) started within the 3 months prior to first dose of study treatment.
* Participants who report treatment with a benzodiazepine, an opioid medication, or a mood stabilizer (such as valproic acid or lithium) within 2 weeks prior to the first dose of esketamine.
* Participants with confirmed psychotic disorder or symptoms, bipolar disorder and or clinically significant alcohol or substance misuse confirmed by a psychiatrist in the previous 2 years.
* Previous ketamine abuse as determined by Investigator
* Previous non-response to clinical or research ketamine administration
* Current diagnosis of bulimia nervosa
* Participants who have been diagnosed with ADD/ADHD and who are also currently taking stimulant medication such as methylphenidate or another amphetamine-type medication.
* Participants currently taking St John's Wort, Ginseng or Turmeric
* Participants judged clinically to be actively at serious risk of self-harm or suicidal behaviour by the study team or psychiatrist at Screening.
* Blood pressure >140/90 at screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery Asberg Depression Rating Scale (MADRS) from screening to Day 28 | Screening, Day 7, 14, 21 and 28
  The MADRS is a clinician rated 10-item scale where individuals score from 0-6 based on the severity of their symptoms, with higher scores indicative of greater severity

SECONDARY OUTCOMES:
Change in Post-traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5) | Screening and Day 28
  A 20-item self-administered measure that assesses the presence and severity of PTSD symptoms. Participants will be asked to rate how bothered they have been by each itme in the past month on a 5-point Likert scale ranging from 0=Not at all to 4 = Extremely. The PCL-5 is easily scored by summing all of the items for a total symptom severity score ranging between 0-80. Clinically meaningful PTSD symptoms are present if items are rated as a minimum of 2 = "Moderate" or higher
Change in Patient Health Questionnaire (PHQ-9) | Screening, Day 2, 5, 9, 12,16, ,19, 23, 26 and 28
  A 9-item self-administered questionnaire to determine the presence and severity of depression which scores each of the 9 DSM-IV criteria as "0" ( not at all), to "3" ( nearly every day).
Change in Generalized Anxiety Disorder Questionnaire (GAD-7) | Screening, Day 2, 5, 9, 12, 16, 19, 23, 26 and 28
  A 7- item self-administered questionnaire to measure the severity of the levels of anxiety. Each item can be score 0-3, giving a total score of 0-21.
Change in Rosenberg Self-Esteem Questionnaire (RSES) | Screening and Day 28
  A 10-item self-administered questionnaire to measure change in self esteem following psychological intervention. Each item scoring from 1-4, and higher scores indicating greater self-esteem
Change in Quality of Life 8 Dimensional Questionnaire (AQoL-8D) | Screening and Day 28
  Self administered questionnaire measuring quality of life across 8 domains: independent living, happiness, mental health, coping, relationships, self-worth, pain and senses.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chue, MBBCh, Principal Investigator — Amygdala Associates
Locations (1):
- City Center Pharmacy and Medical Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other members of the research team including Dr. Craig Buchholz
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Throughout the study.
Access Criteria: Involved in data collection